CLINICAL TRIAL: NCT06159842
Title: An Investigator Initiated Study to Evaluate the Safety and Efficacy of Aminolevulinic Acid 20% Topical Solution (Levulan® Kerastick®) (ALA) + Blue Light in the Treatment of Facial Cutaneous Squamous Cell Carcinoma in Situ (isSCC)
Brief Title: Evaluating the Use of Photodynamic Therapy to Treat Facial Cutaneous Squamous Cell Carcinoma in Situ (isSCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Center for Clinical and Cosmetic Research (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Principal Investigator, Mark Steven Nestor, M.D., Ph.D., Director, The Center for Clinical and Cosmetic Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCCR 03-2023
Record Dates: First submitted 2023-11-20; First posted 2023-12-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-08

CONDITIONS: Facial Cutaneous Squamous Cell Carcinoma in Situ
Keywords: skin cancer; facial skin cancer; Squamous Cell Carcinoma; Squamous Cell Carcinoma in Situ; Cutaneous Squamous Cell Carcinoma in Situ; Facial Cutaneous Squamous Cell Carcinoma in Situ
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Squamous Cell; Squamous Intraepithelial Lesions | interventions — Aminolevulinic Acid; Solutions; Blue Light

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Photodynamic Therapy (Blue light dose 10 J/cm2 at 10 mW/cm2) (Experimental): 30 participants will be enrolled to this arm
  Interventions: Combination Product: Aminolevulinic Acid 20% Topical Solution with Blue Light

INTERVENTIONS:
Combination Product: Aminolevulinic Acid 20% Topical Solution with Blue Light — Participants will have their facial isSCC prepped then treated with Aminolevulinic Acid 20% Topical Solution (Levulan® Kerastick® Applicators) (ALA), followed by blue light therapy administered for 16 minutes and 40 seconds to deliver the total desired light dose to the isSCC lesion.
  Other Names: Levulan® Kerastick®; BLU-U® Blue Light Photodynamic Therapy Illuminator

SUMMARY:
The goal of this clinical trial is to test how safe and effective it is to treat early form of cancer cells found in the upper skin layer of the face, using a light-sensitive cream used in combination with a light source.

The main questions this trial aims to answer are:

* to confirm using laboratory testing, how much of the affected facial skin cancer section the treatment was able to remove, and;
* seeing how many participants had no remaining affected facial skin cancer sections after treatment.

Participants who qualify will be asked to complete 12 visits in total and will receive a total of two treatments, after voluntarily consent has been given.

DETAILED DESCRIPTION:
In the study, participants will be asked to complete the following:

* Provide basic personal information (including date of birth, gender, race and ethnicity)
* Provide their medical/ surgical history and perform a medical exam (including but not limited to physical exam, skin type, vital signs, height, weight and urine pregnancy test collection)
* Follow study rules such as avoiding certain medications and treatments
* Allow photographs of the area of skin cancer being treated on the face
* Provide information on any medications, treatments or reactions that started after the study began
* Allow two treatments on the skin cancer area of the face using a light-sensitive cream used in combination with a light source
* Allow clinical documentation of the treatment, such as how well the treatment was tolerated, any skin reaction or side effects
* Allow surgery to remove the skin cancer area from the face for Laboratory testing

To qualify for this trial, participants must:

* be an adult (18 years of age or older)
* give voluntary written consent
* have a recently diagnosed (less than six months from first visit) skin cancer area on the face that meets surgery size requirements
* be willing to follow study instructions and complete study requirements, including not using non-approved lotions and creams on the treatments areas
* (if female) not be pregnant before and during the study and agree to use acceptable forms of birth control
* confirm they are not sensitive to any of the study treatment ingredients

All surgery samples collected from the participants towards the end of the study will be sent to a laboratory for testing. All photographs of the treatment area collected during the study will be used as study data.

All participants have the right to refuse further participation in the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Must be an adult (18 years of age or older)
* Voluntary written consent required
* Must have a recently diagnosed (no more than six months from first study visit) facial isSCC lesion that meets surgery excision size requirements
* Cannot have other dermatological disease in the isSCC target area
* Must be willing to follow study instructions and complete study requirements, including not using non-approved lotions and creams on the treatments areas
* If female, cannot be pregnant before and during the study and agree to use acceptable forms of birth control

Exclusion Criteria:

* Sensitive to any of the study treatment ingredients
* Pregnant or lactating
* Medical laboratory evidence of other non-isSCC tumor in the target lesion biopsy specimen
* History of recurrence in the target isSCC lesion
* Medical laboratory evidence of certain growth patterns in the target lesion biopsy specimen
* Chronic medical condition that in the Investigators opinion will interfere in the trial or affect participant safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with Histological Clearance of treated isSCC lesion | Up to 16 weeks
  Histological clearance is defined as the absence of detectable evidence of isSCC tumor cell nests by the central pathology reports

SECONDARY OUTCOMES:
Number of participants with clinical clearance of treated isSCC lesion | through treatment completion, an average of 12 weeks
  Complete Clinical Clearance will be measured by the Investigator and is defined as when there is no clinically visible lesion remaining at the site.
Local Skin Response Scale | up to 16 weeks
  Observations and changes noted in the aesthetic appearance (Erythema, Flaking/ Scaling, Crusting, Swelling, Vesiculation/ Pustulation, Erosion/ Ulceration) of the treated isSCC lesion will each be graded on a scale of 0 to 4, with 0 as no presence and 4 as a severe outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nestor, MD, PhD, Principal Investigator — Center for Clinical and Cosmetic Research
Locations (1):
- Center for Clinical and Cosmetic Research, Aventura, Florida, United States